CLINICAL TRIAL: NCT03500094
Title: An Open-label Study of the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of 12 Month Treatment With Migalastat in Pediatric Subjects (Aged 12 to <18 Years) With Fabry Disease and Amenable GLA Variants
Brief Title: Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of Migalastat in Pediatric Subjects (Aged 12 to <18 Years)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT1001-020; 2017-000146-21 (EudraCT Number)
Expanded Access: NCT01476163 (Available)
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Results first posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Fabry Disease
Keywords: Lysosomal storage disease; migalastat; AT1001; Galafold
MeSH Terms: conditions — Fabry Disease; Lysosomal Storage Diseases | interventions — migalastat; larazotide acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- migalastat HCl 150 mg (Experimental): One migalastat 123 milligrams (mg) capsule equivalent to 150 mg migalastat hydrochloride (HCl) (herein referred to as "migalastat") was administered every other day for 12 months.
  Interventions: Drug: Migalastat HCl 150 mg

INTERVENTIONS:
Drug: Migalastat HCl 150 mg — migalastat HCl 150 mg capsule
  Other Names: AT1001; Galafold

SUMMARY:
This was an open-label study to evaluate the safety, pharmacokinetics (PK), pharmacodynamics (PD), and efficacy of migalastat treatment in pediatric participants 12 to <18 years of age with Fabry disease and amenable gene encoding α-galactosidase A (GLA) variants.

DETAILED DESCRIPTION:
This was a Phase 3b, 2-stage, open-label, uncontrolled, multicenter study to evaluate the safety, PK, PD, and efficacy of migalastat treatment in pediatric participants 12 to <18 years of age and weighing ≥ 45 kilograms (99 pounds) with Fabry disease and amenable GLA variants. Participants must have been naïve to enzyme replacement therapy (ERT) or have stopped ERT at least 14 days at the time of screening.

Stage 1 was a treatment period of approximately 1 month (4 weeks); Stage 2 was a treatment period of 11 months and a 30-day (untreated) safety follow-up period. There was no break in treatment between Stages 1 and 2. Prior to Stage 1, there was a screening period lasting at least 14 days and up to 30 days (or more, if GLA genotyping was required). Stages 1 and 2 together consisted of a 12-month treatment period, and a 30-day safety follow-up period, for a total of approximately 13 months. Upon study completion, participants had the option to enroll in a long-term extension study conducted under a separate protocol (NCT04049760).

Participants were randomly assigned 1:1:1 to 1 of 3 PK sampling groups using interactive response technology (IRT). Four blood samples for the determination of migalastat concentrations in plasma were collected during Stage 1 study drug administration, and 1 PK (trough) sample was collected at Month 6 and again at Month 12.

ELIGIBILITY:
Key Inclusion Criteria

* Willing and able to provide written consent or assent (participant and parent/legal guardian, as applicable)
* Male or female between 12 and <18 years of age diagnosed with Fabry disease
* Confirmed, amenable GLA variant
* Participant weighed at least 45 kg (99 pounds) at screening
* Participant had never been treated with ERT or had not received ERT for 14 days prior to screening
* Participant had at least 1 complication (such as, laboratory abnormality and/or sign/symptom) of Fabry disease
* Participant was able to swallow study medication whole

Key Exclusion Criteria

* Had moderate or severe renal impairment (estimated glomerular filtration rate (eGFR) <60 milliliter/minute/1.73 meter squared (m^2) at screening)
* Had advanced kidney disease requiring dialysis or kidney transplantation
* History of allergy or sensitivity to study medication (including excipients) or other iminosugars (for example, miglustat, miglitol)
* Had received any gene therapy at any time or anticipated starting gene therapy during the study period
* Required treatment with Glyset (miglitol) and/or Zavesca (miglustat) within 6 months before screening or throughout the study
* Required treatment with Replagal (agalsidase alfa), or Fabrazyme (agalsidase beta) within 14 days before screening or throughout the study
* Participant was treated or had been treated with any investigational/experimental drug, biologic or device within 30 days before screening
* Any intercurrent illness or condition or concomitant medication use considered to be a contraindication at screening or baseline or that may have precluded the participant from fulfilling the protocol requirements or suggested to the investigator that the potential participant may have had an unacceptable risk by participating in this study
* Pregnant or breast-feeding or planned to become pregnant during the study period
* Otherwise unsuitable for the study in the opinion of the investigator

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor Clinical Research, Study Director — Amicus Therapeutics
Locations (8):
- United States (7):
  - Clinical Study Site, Tampa, Florida
  - Clinical Study Site, Atlanta, Georgia
  - Clinical Study Site, Minneapolis, Minnesota
  - Clinical Study Site, Columbia, Missouri
  - Clinical Study Site, Cincinnati, Ohio
  - Clinical Study Site, Pittsburgh, Pennsylvania
  - Clinical Study Site, Fairfax, Virginia
- Clinical Study Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants must have been either naïve to enzyme replacement therapy (ERT) or have stopped ERT at least 14 days at the time of screening.
Groups:
- Migalastat HCl 150 mg: Migalastat was administered every other day for 12 months.
Period: Overall Study
Arm/Group | Migalastat HCl 150 mg
Started | 22
Received At Least 1 Dose of Study Drug | 21
Completed | 19
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Withdrawal by Parent or Legally-authorized Representative | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: All participants who enrolled in the study.
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.6 (1.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 10
Race/Ethnicity, Customized [Number; unit: participants]
  White | 20
  Other | 2
  Hispanic or Latino | 3
  Not Hispanic or Latino | 19

OUTCOME MEASURES:

1. Primary Outcome: Number Of Participants Who Experienced Treatment-related Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs included adverse events that began on or after the first dose of study drug until 30 days after the last dose. Treatment-related TEAEs were defined as TEAEs that had an investigator-defined relationship to study drug of "Definite," "Probable," or "Possible." A summary of serious and all other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Day 1 (after dosing) through Month 12 and follow-up (30 days after last dose)
Population: Participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 21
Participants | 5

2. Primary Outcome: Pharmacokinetics (PK): Area Under The Plasma Concentration-time Curve Over The Dosing Interval (AUCtau) Of Migalastat
Description: PK sampling was performed on 1 occasion at steady-state during the first month of the study. Adolescent participants were randomized to 3 sparse PK sampling groups based on optimal sampling theory. Each blood sample could have been taken at any time within the following time point ranges. Time point ranges for all 3 sparse sampling groups are arranged here in chronological order: 1 to 1.25 hours (h), 1.5 to 2h, 2.75 to 3.25h, 3.25 to 3.75h, 3.75 to 4.25h, 5 to 5.5h, 5.25 to 5.75h, 6.5 to 7h, 8.25 to 8.75h, 8.75 to 9.25h, and 10.75 to 11.25h post-dose. The combined sampling scheme resulted in rich data over an approximate 12-hour time course for AUC estimation. Additional trough samples were taken at Months 6 and 12. These trough samples (48h) assisted in estimating the terminal elimination phase for the AUC.
  Simulations were conducted to predict steady-state PK profiles and parameters for adolescent age subgroups 12 to <16 years, 16 to <18 years, and overall, 12 to <18 years.
Time Frame: 0 to 12 hours postdose during the first month of study and trough samples at Months 6 and 12
Population: Participants with at least 1 quantifiable concentration and a known weight and estimated glomerular filtration rate (eGFR). A population PK model was used for assessment. All migalastat concentration-time data were combined and included in a population PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 20
h*ng/mL
  12 to <16 years old: number analyzed (Participants) | 13
  12 to <16 years old | 8920 (47.2)
  16 to <18 years old: number analyzed (Participants) | 7
  16 to <18 years old | 8430 (41.7)
  12 to <18 years old | 8740 (44.2)

3. Primary Outcome: PK: Maximum Observed Plasma Concentration (Cmax) Of Migalastat
Description: PK sampling was performed on 1 occasion at steady-state during the first month of the study. Adolescent participants were randomized to 3 sparse PK sampling groups based on optimal sampling theory. Each blood sample could have been taken at any time within the following time point ranges. Time point ranges for all 3 sparse sampling groups are arranged here in chronological order: 1 to 1.25h, 1.5 to 2h, 2.75 to 3.25h, 3.25 to 3.75h, 3.75 to 4.25h, 5 to 5.5h, 5.25 to 5.75h, 6.5 to 7h, 8.25 to 8.75h, 8.75 to 9.25h, and 10.75 to 11.25h post-dose. The combined sampling scheme resulted in rich data over an approximate 12-hour time course for AUC and Cmax estimation. Additional trough samples were taken at Months 6 and 12. These trough samples (48h) assisted in estimating the terminal elimination phase for the AUC.
  Simulations were conducted to predict steady-state PK profiles and parameters for adolescent age subgroups 12 to <16 years, 16 to <18 years, and overall, 12 to <18 years.
Time Frame: 0 to 12 hours postdose during the first month of study and trough samples at Months 6 and 12
Population: Participants with at least 1 quantifiable concentration and a known weight and eGFR. A population PK model was used for assessment. All migalastat concentration-time data were combined and included in a population PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 20
ng/mL
  12 to <16 years old: number analyzed (Participants) | 13
  12 to <16 years old | 1220 (60.9)
  16 to <18 years old: number analyzed (Participants) | 7
  16 to <18 years old | 1160 (39.2)
  12 to <18 years old | 1200 (52.7)

4. Secondary Outcome: Change In eGFR From Baseline To Month 12
Description: eGFR was calculated using the modified Schwartz formula for creatinine clearance.
Time Frame: Baseline, Month 12 and last observation (up to Month 12)
Population: Participants who received at least 1 dose of study drug and had evaluable data at the specified timepoints.
Measure: Mean (Standard Deviation); unit: mL/min x 1.73 m^2
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 20
mL/min x 1.73 m^2
  Month 12: number analyzed (Participants) | 19
  Month 12 | -1.6 (15.40)
  Last observation (up to Month 12) | -1.6 (14.99)

5. Secondary Outcome: Annualized Rate Of Change From Baseline
Description: Annualized rate of change from baseline of eGFR was defined as change from baseline to last visit divided by the duration from baseline to the last visit (Last assessment date - First dose date +1) and multiplied by 365.25. Baseline was defined as the last non-missing assessment prior to the first dose of study drug.
Time Frame: Baseline up to Month 12
Population: All participants who received study drug and had an assessment
Measure: Mean (Standard Deviation); unit: mL/min x 1.73 m^2/year
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 20
mL/min x 1.73 m^2/year | -1.5 (15.11)

6. Secondary Outcome: Change From Baseline In Total Urine Protein And Urine Albumin Levels At Month 12
Description: Renal function was assessed by urine protein and urine albumin levels. Urine samples were collected as part of urinalysis to measure protein and albumin levels.
Time Frame: Baseline, Month 12 and last observation (up to Month 12)
Population: Participants who received at least 1 dose of study drug and had evaluable data at the specified timepoints.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 20
mg/L
  Total Urine Protein: Month 12: number analyzed (Participants) | 19
  Total Urine Protein: Month 12 | 36.0 (111.61)
  Total Urine Protein: Last observation (up to Month 12) | 36.2 (108.64)
  Urine Albumin: Month 12: number analyzed (Participants) | 19
  Urine Albumin: Month 12 | 16.2 (28.27)
  Urine Albumin: Last observation (up to Month 12) | 15.6 (27.67)

7. Secondary Outcome: Change From Baseline In Left Ventricular Mass Index (LVMi)
Description: LVMi was assessed as a measure of cardiac impairment in the study participants. LVMi values for both M Mode and 2D views are presented.
Time Frame: Baseline, Month 12 and last observation (up to Month 12)
Population: Participants who received at least 1 dose of study drug and had evaluable data at the specified timepoints.
Measure: Mean (Standard Deviation); unit: g/m^2
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 20
g/m^2
  M Mode: Month 12: number analyzed (Participants) | 18
  M Mode: Month 12 | -3.9 (13.53)
  2D: Month 12: number analyzed (Participants) | 19
  2D: Month 12 | 4.9 (9.12)
  M Mode: Last observation (up to Month 12): number analyzed (Participants) | 19
  M Mode: Last observation (up to Month 12) | -4.4 (13.31)
  2D: Last observation (up to Month 12) | 4.3 (9.34)

8. Secondary Outcome: Change In Plasma Levels Of Globotriaosylsphingosine (Lyso-Gb3)
Description: Blood samples were collected for measurement of lyso-Gb3 levels in plasma. Plasma levels of lyso-Gb3 were measured using a validated liquid chromatography-mass spectrometry assay.
Time Frame: Baseline, Month 12 and last observation (up to Month 12)
Population: Participants who received at least 1 dose of study drug and had evaluable data at the specified timepoints.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Migalastat HCl 150 mg: ERT Naive: Migalastat was administered every other day for 12 months to ERT Naive participants.
- Migalastat HCl 150 mg: ERT Experienced: Migalastat was administered every other day for 12 months to ERT experienced participants.
Arm/Group | Migalastat HCl 150 mg: ERT Naive | Migalastat HCl 150 mg: ERT Experienced
Number analyzed (Participants) | 9 | 11
ng/mL
  Month 12: number analyzed (Participants) | 9 | 10
  Month 12 | -14.0 (23.13) | 12.5 (36.33)
  Last Observation (up to Month 12) | -14.0 (23.13) | 11.3 (34.67)

9. Secondary Outcome: FABPRO-GI And Pain Scores
Description: The Fabry Disease Patient-Reported Outcome - Gastrointestinal Signs And Symptoms (FABPRO-GI) And Pain Questionnaire For Clinical Trials (24-hr Version) consists of questions regarding gastrointestinal signs and symptoms and pain relative to the past 24 hours. Participants rated the severity of their symptoms and pain from 0 (none) to 10 (worst possible). The monthly average score at Month 12 and at last observation are presented. A higher score indicated higher levels of symptoms and pain.
Time Frame: Month 12 and last observation (up to Month 12)
Population: Participants who received at least 1 dose of study drug and had evaluable data at the specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 18
units on a scale
  Daily Ratings of Severity in Constipation: Month 12: number analyzed (Participants) | 5
  Daily Ratings of Severity in Constipation: Month 12 | 0.9 (1.91)
  Daily Ratings of Severity in Constipation: Last observation (up to Month 12) | 0.4 (1.00)
  Daily Ratings of Severity in Diarrhea: Month 12: number analyzed (Participants) | 5
  Daily Ratings of Severity in Diarrhea: Month 12 | 1.0 (1.65)
  Daily Ratings of Severity in Diarrhea: Last Observation (up to Month 12) | 0.4 (0.91)
  Overall Pain: Month 12: number analyzed (Participants) | 5
  Overall Pain: Month 12 | 0.6 (0.71)
  Overall Pain: Last Observation (up to Month 12) | 1.2 (1.50)
  Worst Tummy Pain: Month 12: number analyzed (Participants) | 5
  Worst Tummy Pain: Month 12 | 0.3 (0.38)
  Worst Tummy Pain: Last Observation (up to Month 12) | 0.9 (1.52)

10. Secondary Outcome: Patient's Global Impression Of Change (PGI-C) Scores
Description: The PGI-C consists of 4 questions regarding diarrhea, abdominal pain, overall pain, and daily living. Participants rated their status based on improvement, worsening, or the same. Improved status includes "Much better", "Better" and "A little better"; worsened status includes "A little worse", "Worse" and "Much worse".
Time Frame: Month 12
Population: Participants who received at least 1 dose of study drug and had evaluable data at the specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 19
Participants
  Diarrhea: Status Improved | 12
  Diarrhea: Status Same | 7
  Diarrhea: Status Worse | 0
  Abdominal pain: Status Improved | 10
  Abdominal pain: Status Same | 8
  Abdominal pain: Status Worse | 1
  Overall pain: Status Improved | 10
  Overall pain: Status Same | 8
  Overall pain: Status Worse | 1
  Daily living: Status Improved | 10
  Daily living: Status Same | 8
  Daily living: Status Worse | 1

11. Secondary Outcome: Number Of Participants Who Experienced Sudden Onset Of Pain As Assessed Using The Fabry-Specific Pediatric Health And Pain Questionnaire (FPHPQ)
Description: The assessment of "In the last 3 months how many times did you experience sudden onset of pain?" using the FPHPQ for ages 13 to 18 is presented.
Time Frame: Month 12
Population: Participants who received at least 1 dose of study drug and had evaluable data at the specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 19
Participants
  0 times | 4
  1-3 times | 5
  4-6 times | 4
  > 6 times | 3

12. Secondary Outcome: Change From Baseline In FPHPQ Score For Pain Intensity
Description: The assessment of "How bad is your pain today?" using the FPHPQ for ages 13 to 18 is presented. Pain intensity was measured on a 10-point scale, 0 (no pain) to 10 (pain as bad as you can imagine). A decrease from baseline indicates an improvement in the condition.
Time Frame: Baseline, Month 12 and last observation (up to Month 12)
Population: Participants who received at least 1 dose of study drug and had evaluable data at the specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 17
units on a scale
  Month 12: number analyzed (Participants) | 16
  Month 12 | 0.4 (1.82)
  Last observation (up to Month 12) | 0.4 (1.77)

13. Secondary Outcome: Change From Baseline In Pediatric Quality Of Life (PedsQL) At Month 12
Description: The PedsQL is a modular approach to measuring health-related quality of life in healthy children and adolescents and those with acute and chronic health conditions. The psychosocial score for the PedsQL encompassed 15 questions relating to the participants' feelings, social interaction with others, and school. The physical score was derived from answers to 8 questions about the participants' ease of managing physical activity.
  All components of the PedsQL were scored based on a scale of 0 (never) to 4 (almost always) and linearly transformed to a 0-100 scale as follows: 0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0. Both categories were combined for a total score. Total scores for the child report ages 13 to 18 years old and parent report are presented at Month 12.
Time Frame: Baseline, Month 12
Population: Participants who received at least 1 dose of study drug and had evaluable data at the specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Migalastat HCl 150 mg
Number analyzed (Participants) | 15
units on a scale
  Child Report | 2.2 (6.13)
  Parent Report | 3.1 (10.29)

ADVERSE EVENTS:
Time Frame: Day 1 (after dosing) through Month 12 and follow-up (30 days after last dose)
Arm/Group | Migalastat HCl 150 mg
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 1/21
Other Adverse Events (participants affected / at risk) | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Migalastat HCl 150 mg (N=21)
Suicidal ideation (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Migalastat HCl 150 mg (N=21)
Vomiting (Gastrointestinal disorders) | 2
Complication associated with device (General disorders) | 2
Influenza (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 3
Pharyngitis streptococcal (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 3
Paraesthesia (Nervous system disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator can publish only the results from this trial, provided they supply the sponsor (or authorized entity) a copy of any proposed publication for review prior to submission for publication. If requested and prior to publication, the investigator will remove information deemed confidential or proprietary by the sponsor and will withhold publication an additional period of time to allow the sponsor to take appropriate measures to establish and preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT03500094/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/94/NCT03500094/SAP_001.pdf